CLINICAL TRIAL: NCT06892392
Title: Aplicación Del ICG En La Linfadenectomía D2 Laparoscópica Del Cáncer Gástrico Localmente Avanzado: Ensayo Clínico Aleatorizado Multicéntrico.
Brief Title: Application of Indocyanine Green Tracer in D2 Lymphadenectomy of Locally Advanced Gastric Cancer
Acronym: Gastri-ICG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital of Navarra (Other)
Responsible Party: Principal Investigator, Ines Eguaras, Principal investigator, Hospital of Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hospital Universitario de Nava
Record Dates: First submitted 2025-03-10; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: GASTRIC CANCER; Indocyanine Green (ICG); Lymph Node Excision; Lymphadenectomy; Laparoscopic Gastrectomy
Keywords: Multicenter randomized 1:1 clinical trial; indocyanine green; Laparoscopic gastrectomy with D2 lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group, Subtotal/Total gastrectomy with D2 lymphadenectomy LPS ( standar of care) (No Intervention): * Tumor localization and assessment of resectability
  * Omentectomy
  * Ligation and dissection of the right gastroepiploic vessels at their origin.
  * Dissection of lymph node group 6
  * Opening of the pars flaccida of the lesser omentum.
  * Dissection and ligation of the pyloric artery at its origin
  * Dissection of ganglionic group 5
  * Dissection and section of the first portion of the duodenum.
  * Lymphadenectomy D2: 7, 8, 9, 9, 11 p, 12a
  * Ligation and section of the coronary artery at origin
  * Group 1 lymphadenectomy
  * Gastric section with negative margin
  * Removal of the specimen
  * Reconstruction according to the usual technique
  Ex vivo analysis of the specimen in the surgical block. A dissection of the D2 lymphadenectomy lymph node groups will be performed including the following groups according to the Japanese Gastric Cancer Association Classification:
  - Group 7, 8, 9, 11 p, 12 a. Each lymph node group will be sent in a separate labeled sample bottle to the pathology department.
- Intervention group: ICG administration (Experimental): ICG administration: For ICG administration, a gastroscopy must be performed by the Digestive Service of each center, with sedation 24 h before surgery. For this, the lesion is located by gastroscopy, after which it is injected in 4 quadrants in the submucosa, with a total volume of 2 ml.
  To prepare the ICG, 0.5 ml (containing 0.625 mg of ICG) is dissolved in 1.25 mg/dl of sterile water
  Standard Total or Subtotal gastrectomy and D2 lymphadenectomy will be performed. After removal of the specimen, we will use ICG mode and evaluate if there are foci of uptake in the territory of the D2 lymphadenectomy.
  - If there are foci of uptake, dissect and resect them. Identified in a separate anatomic pathology jar and labeled with the name of the corresponding anatomic region with ICG
  Interventions: Procedure: ICG administration

INTERVENTIONS:
Procedure: ICG administration — For the administration of ICG, it is necessary to perform a gastroscopy by the Digestive Service of each center, with sedation 24 h before surgery. For this, the lesion is located by gastroscopy, after which it is injected in 4 quadrants in the submucosa, with a total volume of 2 ml.
  To prepare the ICG, 0.5 ml (containing 0.625 mg of ICG) is dissolved in 1.25 mg/dl of sterile water
  Other Names: ICG
  Arms: Intervention group: ICG administration

SUMMARY:
Gastric cancer is a frequent neoplasm in the world, presenting more than one million new cases and around 768,000 deaths in the data registered in 2020. Among the therapeutic options for gastric cancer, surgery is an essential pillar for its treatment. Gastric cancer surgery consists of gastric resection with negative margins and radical lymphadenectomy in patients without distant metastases. It has been demonstrated over the years that radical lymphadenectomy in gastric cancer allows for adequate staging and improved long-term survival.

In order to perform a correct staging using the TNM system, it is necessary to resect at least 15 lymph nodes in the radical lymphadenectomy. For radical lymphadenectomy staging, the Japanese Gastric Cancer Association defined and subdivided nodal stations. Three types of lymphadenectomy are described according to oncologic gastric resections (D1, D1+ and D2), with D2 lymphadenectomy being the standard of treatment for locally advanced gastric tumors. Performing an insufficient or inadequate lymphadenectomy has been shown to negatively impact survival after gastrectomy in such a cohort.

The development of technology based on fluorescence guided by indocyanine green could improve the technique and results of D2 lymphadenectomy in patients with gastric cancer. There is evidence that the application of ICG in D2 lymphadenectomy increases the number of resected nodes, however, studies of higher scientific quality (randomized clinical trials) are needed. Furthermore, most studies in this field have focused on Eastern countries (Japan, Korea and China), where the percentage of early tumors and chemotherapy treatment is different from Western centers.

Therefore, we propose a multicenter randomized clinical trial aimed at evaluating whether the application of ICG-guided fluorescence-based technology in D2 lymphadenectomy of locally advanced gastric cancer increases the number of resected nodes, improves the oncologic quality of the lymphadenectomy, and thus may increase overall survival and disease-free survival at 2 and 5 years postoperatively.

DETAILED DESCRIPTION:
Objective:

- Mean total number of nodes/ nodal ratio (number of positive nodes divided by the number of total nodes).

Secondary objective:

* Overall Survival and disease- free survival at 2 and 5 years.
* Number of metastatic nodes
* Complications measured with the Comprehensive Complication Index (CCI)
* Intraoperative bleeding volume
* Surgical time (minutes)
* Days of hospitalization (days) Randomized clinical trial 1:1. The patient will be included once the perioperative chemotherapy treatment is completed. The investigator at each center will explain the study, and if the patient consents to participate, he/she will sign the informed consent form (IC). After which, the investigator of each center will contact the principal investigator of the University Hospital of Navarra (HUN), who will perform the randomization and communicate the result by email to the participating center.

Requirements for participating centers:

* Esophagogastric Surgery Unit with a volume of 20 patients with gastric neoplasia operated on in one year.
* Use the 4k Rubina Tower of the Karl Storz brand.

Inclusion criteria:

* < 85 years
* T1/T4a, N+, M0 in the preoperative study.
* PS 0-1
* ASA I-III
* Laparoscopic surgery

Exclusion criteria:

* Previous gastric abdominal surgery
* DSE
* Cognitive impairment
* Allergic to iodine
* Synchronous neoplasm
* Stroke in the last 6 months
* Angina or AMI in the last 6 months
* Plastic lymphitis
* Open surgery

ICG administration: For ICG administration, a gastroscopy must be performed by the Digestive Service of each center, with sedation 24 hours before surgery. For this, the lesion is located by gastroscopy, after which it is injected in 4 quadrants in the submucosa, with a total volume of 2 ml.

To prepare the ICG, 0.5 ml (containing 0.625 mg of ICG) is dissolved in 1.25 mg/dl of sterile water.

ELIGIBILITY:
Inclusion Criteria:

* T2-T4a, N+, M0 on preoperative study
* PS 0-1
* ASA I-III
* Laparoscopic surgery

Exclusion Criteria:

* - Previous gastric abdominal surgery
* DSE
* Cognitive impairment
* Allergic to iodine
* Synchronous neoplasm
* Stroke in the last 6 months
* Angina or AMI in the last 6 months
* Plastic lymphitis
* Open surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
total nodes resected | 18 months
  Mean of the total nodes resected in the D2 lymphadenectomy
Nodal ratio | 18 months
  number of positive nodes divided by number of total nodes

SECONDARY OUTCOMES:
Overall Survival | 2 and 5 years
  Overall survival at 2 and 5 years
Disease-free survival | 2 and 5 years
  Disease-free survival at 2 and 5 years
Number of metastatic nodes | 18 months
  Number of metastatic nodes
Comprehensive Complication Index | 30 days after surgery
  Comprehensive Complication Index (CCI)
Intraoperative bleeding volume | 18 months
  Intraoperative bleeding volume (ml)
Surgical time | 18 months
  Surgical time (minutes)
Days of hospitalization | 18 months
  Days of hospitalization
Correlation of positive lymph nodes in anatomical pathology and with ICG uptake | 18 months
  Correlation of positive lymph nodes in anatomical pathology and with ICG uptake

CONTACTS AND LOCATIONS:
Overall Officials: Maria Concepcion Yarnoz, MD, PhD, Study Chair — Hospital of Navarra
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No